CLINICAL TRIAL: NCT01309945
Title: A Multicenter, Randomized, Double-blind, Active-Controlled Study of the Efficacy and Safety of Flexibly-Dosed BMS-820836 in Patients With Treatment Resistant Major Depression
Brief Title: Efficacy and Safety of Flexibly Dosed BMS-820836 in the Treatment of Patients With Treatment Resistant Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN162-006; 2010-022841-93 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-03-07 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride; 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1: Duloxetine 30mg (Active Comparator)
  Interventions: Drug: Duloxetine
- Arm 2: BMS-820836 placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching with BMS-820836
- Arm 3: BMS-820836 0.5-2.0 mg/day (Experimental)
  Interventions: Drug: BMS-820836
- Arm 4: Duloxetine 30mg (Active Comparator)
  Interventions: Drug: Duloxetine
- Arm 5: Duloxetine placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching with Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Capsule, Oral, 30-60 mg/day, once daily (QD), 8 weeks
  Other Names: Cymbalta
  Arms: Arm 1: Duloxetine 30mg
Drug: Placebo matching with BMS-820836 — Tablet, Oral, 0.0 mg, once daily (QD), 14 weeks
  Arms: Arm 2: BMS-820836 placebo
Drug: BMS-820836 — Tablet, Oral, 0.5-2.0 mg, once daily (QD), 6 weeks
  Arms: Arm 3: BMS-820836 0.5-2.0 mg/day
Drug: Duloxetine — Capsule, Oral, 30-60 mg/day, once daily (QD), 6 weeks
  Other Names: Cymbalta
  Arms: Arm 4: Duloxetine 30mg
Drug: Placebo matching with Duloxetine — Tablet, Oral, 0.0 mg, once daily (QD), 8 weeks
  Arms: Arm 5: Duloxetine placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of study drug (BMS-820836) as compared with continued duloxetine in the treatment of patients with treatment resistant depression (TRD).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use.
* Patients with a diagnosis of Major Depressive Disorder, currently experiencing a Major Depressive Episode, as defined by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition Text Revision(DSM IV TR) criteria. The current depressive episode must be > 8 weeks in duration and < 3 years duration.
* In the current Major Depressive Disorder (MDD) episode, patients should report a history of inadequate response to 1 - 3 adequate trials of antidepressant treatment.
* Patients must have a 17-item Hamilton Depression Rating Scale (HAM-D17) total score =>18 at Screening.

Exclusion Criteria:

* Patients who report an inadequate response (less than 50% reduction in depressive symptom severity) to more than three adequate trials of antidepressant treatments during the current depressive episode.
* Patients who have failed duloxetine at an adequate dose and for an adequate duration in their current episode unless in the judgment of the investigator, the patient could benefit from the treatment with this medication.
* Patients whose only inadequate response to an antidepressant in the current Major Depressive Episode (MDE) is to an Serotonin norepinephrine reuptake inhibitors (SNRI) (duloxetine, venlafaxine, desvenlafaxine or milnacipran).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) total score | End of phase B and End of phase C

SECONDARY OUTCOMES:
Change in Sheehan Disability Scale (SDS) Total score | End of Phase B and End of Phase C
Change in the Montgomery Asberg Depression Rating Scale (MADRS) anhedonia factor score | End of Phase B and End of Phase C

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (83):
- United States (55):
  - K & S Professional Research Services, Llc, Little Rock, Arkansas
  - Pacific Clinical Research Medical Group, Arcadia, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - California Neuropsychopharmacology Clinical Research Inst., San Diego, California
  - Pacific Research Network, Inc, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Radiant Research, Inc., Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, Llc, Orlando, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Atlanta Institute Of Medicine & Research, Atlanta, Georgia
  - Comprehensive Clinical Development, Inc., Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Loyola University Health System, Maywood, Illinois
  - Alpine Clinic, Lafayette, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - James G. Barbee, Md, Llc, New Orleans, Louisiana
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richard H. Weisler, Md, Pa & Assoc., Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Ips Research Company, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Oregon Center For Clinical Investigations, Inc. (Occi, Inc), Portland, Oregon
  - Summit Research Network (Oregon) Inc, Portland, Oregon
  - Oregon Center For Clinical Investigations, Inc (Occi, Inc), Salem, Oregon
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Univ Of Penn, Philadelphia, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Belmont Center For Comprehensive Treatment, Philadelphia, Pennsylvania
  - University Of Pennsylvania, Philadephia, Pennsylvania
  - Carolina Clinical Research Services, Columbia, South Carolina
  - University Of South Carolina School Of Medicine, Columbia, South Carolina
  - Psychiatric Consultants, Pc, Franklin, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - Uthealth - Houston, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - San Antonio Psychiatric Research Center, San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - Psychiatric And Behavioral Solutions, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) Llc, Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin
  - Independent Psychiatric Consultants, Sc, Dba, Ipc Research, Waukesha, Wisconsin
- Canada (5):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Finland (6):
  - Local Institution, Helsinki
  - Local Institution, Jarvenpaa
  - Local Institution, Oulu
  - Local Institution, Seinäjoki
  - Local Institution, Tampere
  - Local Institution, Turku
- France (7):
  - Local Institution, Montpellier, France
  - Local Institution, Nîmes, France
  - Local Institution, Paris, France
  - Local Institution, Dole
  - Local Institution, Douai
  - Local Institution, Élancourt
  - Local Institution, Limoges
- South Africa (6):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Vereeniging, Gauteng
  - Local Institution, Bellville, Western Cape
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Somerset West, Western Cape
- Sweden (4):
  - Local Institution, Halmstad
  - Local Institution, Kungens Kurva
  - Local Institution, Lund
  - Local Institution, Uppsala

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx